CLINICAL TRIAL: NCT01225042
Title: The Effect of Probiotics on E. Coli Gastroenteritis
Acronym: PRETEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N132716.081.10
Record Dates: First submitted 2010-10-15; First posted 2010-10-20 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Gastroenteritis; Bacterial Infection; Diarrhea
Keywords: infectious diarrhea; probiotics; prevention; dietary intervention; E. coli infection; intestinal infection; intestinal resistance
MeSH Terms: conditions — Gastroenteritis; Bacterial Infections; Diarrhea; Dysentery; Escherichia coli Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotics (Experimental): Freeze-dried powder, dose 10E9 CFU twice daily for 4 weeks
  Interventions: Dietary Supplement: probiotics
- placebo (Placebo Comparator): Carrier material powder of identical appearance
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotics — Freeze-dried powder, dose 10E9 CFU twice daily for 4 weeks
  Arms: probiotics
Dietary Supplement: placebo — placebo consisting of carrier material powder of identical appearance
  Arms: placebo

SUMMARY:
Background:

The incidence of gastrointestinal infections is very high. In European countries 10-25% of the population suffers from at least one foodborne infection per year. Probiotics may strengthen human resistance to gut infections as they may beneficially modulate the intestinal microbiota composition and activity, and the immune function upon intestinal infection.

Aim:

To study whether probiotics improve the resistance of humans to enterotoxigenic E. coli (ETEC).

Study design:

The PRETEC study is a parallel, double-blind, placebo-controled 4-weeks intervention with probiotics in healthy volunteers. In this study, the effect of probiotic intervention vs placebo on several infection markers in response to an ETEC challenge is investigated. Participants will be randomly assigned to the probiotic or placebo group (n=21 per group). Subjects will be instructed to maintain their habitual food intake, but to standardize their dietary calcium intake. After an adaptation period of 2 weeks, subjects will be orally infected with a live, but attenuated, ETEC vaccine (strain E1392-75-2A; collection NIZO food research; dose will be 10E10 CFU). This ETEC strain induces mild and short-lived infectious diarrhea symptoms. Before and after infection, a diary will be kept to write down all food and drinks consumption (2x2 days) to assess the habitual dietary intake. The diary will also be used for daily recording of bowel habits and frequency and severity of gastrointestinal complaints. Blood is sampled for immune response analyses and multiple faecal samples are collected to quantify several infection- and immune system markers, to determine probiotic excretion, and to verify dietary calcium intake.

Study population:

Healthy males of 20-55 yrs of age.

Interventions:

Probiotics (freeze-dried powder, dose 10E9 CFU twice daily) or placebo (carrier material powder of identical appearance).

Primary outcomes:

Total fecal ETEC excretion per day and severity of diarrhea (quantified by faecal output per day).

Secondary outcomes:

Serum immune response to ETEC, self-reported stool consistency scores and gastrointestinal complaints, relative faecal wet weight, sIgA and calprotectin in faeces, probiotic persistence and levels of opportunistic pathogens in the endogenous microbiota.

DETAILED DESCRIPTION:
The timeframes for analysis of the primary and secondary outcomes is mentioned below in the Outcome Measures section.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male
* Age 20-55 yrs
* Willingness to replace habitual dairy product intake with the supplied low- calcium soy milk products
* Willingness to abstain from products with high amounts of prebiotic fibers and products with probiotics (except for the supplied one)

Exclusion Criteria:

* Current or previous underlying disease of the GI tract
* lactose intolerance
* Use of antibiotics, norit, laxatives, cholestyramine, acid burn inhibitors, immune suppressiva, prebiotics, probiotics
* detectable serum antibodies against ETEC
* carriage of streptomycin-resistant E. coli in faeces (only relevant when culturing technique for ETEC will be applied instead of specific RT-PCR)
* vegetarians
* heavy alcohol use
* drug use

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Total daily faecal ETEC excretion with time | 1-2 days before ETEC infection and on days 1, 2, 3, 5 and 15 after ETEC infection
Total daily faecal output with time | 1-2 days before ETEC infection and on days 1, 2, 3, 5, 15 after ETEC infection

SECONDARY OUTCOMES:
Bowel habits | Scored daily in a diary
Frequency and severity of gastrointestinal symptoms | Scored daily by VAS scales in a diary
Diarrhea severity | 1-2 days before ETEC infection and on days 1, 2, 3, 5, and 15 after ETEC infection
  Determined as % faecal wet weight
Opportunistic pathogens in faeces | At a single day just before ETEC infection and at a single time point in the first week after ETEC infection
Faecal calprotectin | 1-2 days before ETEC infection and on days 1, 2, 3, 5, and 15 after ETEC infection
Serum antibody response to CFA II | At screening (baseline) and at days 9 and 15 after ETEC infection
Total faecal sIgA | 1-2 days before ETEC infection and on days 1, 2, 3, 5, and 15 after ETEC infection

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Bovee-Oudenhoven, PhD, Principal Investigator — NIZO Food Research; Sandra ten Bruggencate, PhD, Principal Investigator — NIZO Food Research; Arthur Ouwehand, PhD, Principal Investigator — Danisco Finland
Locations (1):
- NIZO food research, Ede, Netherlands

REFERENCES:
- [Result] Ouwehand AC, ten Bruggencate SJ, Schonewille AJ, Alhoniemi E, Forssten SD, Bovee-Oudenhoven IM. Lactobacillus acidophilus supplementation in human subjects and their resistance to enterotoxigenic Escherichia coli infection. Br J Nutr. 2014 Feb;111(3):465-73. doi: 10.1017/S0007114513002547. Epub 2013 Aug 12. PMID 23930950